CLINICAL TRIAL: NCT07312812
Title: The Effect of Art-Based Mandala Coloring Activity on Postpartum Anxiety and Postpartum Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Cahide Çevik, Public health Nursing, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AFYON-HSU-MANDALA-2025
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Depression; Postpartum Anxiety
Keywords: woman; postpartum; depression; anxiety; mandala
MeSH Terms: conditions — Depression, Postpartum; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel-group interventional design. Eligible postpartum women are randomly assigned to either an intervention group or a control group using a lottery-based randomization method. The two groups are followed concurrently throughout the study period without crossover between groups. Participants in the intervention group receive a structured, art-based mandala coloring intervention in addition to routine postpartum care, while participants in the control group receive routine postpartum care only. Outcomes are assessed at multiple predefined time points to evaluate changes over time and to compare the effects of the intervention between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Coloring Activity Group (Experimental): Women who agree to participate in the study will receive individual mandala coloring training by the researcher before hospital discharge. The training will last approximately 20 minutes and will consist of three stages. In the first stage, participants will be informed about mandala coloring. In the second stage, an assistant researcher will demonstrate the coloring process using a sample mandala. The participant will then perform a brief practice on a small sample mandala. In the third stage, a mandala coloring set will be provided for participants to use at home.
  Following the training, participants will be followed for eight weeks with weekly telephone contacts. The first telephone contact will take place during the first week. During this contact, the personal information form and the postpartum anxiety and postpartum depression scales will be administered to collect baseline data. In subsequent contacts, the frequency and duration of mandala coloring activities will be assessed
  Interventions: Behavioral: Mandala Coloring Activity
- Standard of care group (No Intervention): Women in the control group will not receive any intervention. However, postpartum anxiety and postpartum depression scales will be administered by telephone at weeks 1, 4, and 8. During the first week, demographic information will also be collected using a personal information form.

INTERVENTIONS:
Behavioral: Mandala Coloring Activity — Structured mandala coloring training and home practice.
  Arms: Mandala Coloring Activity Group

SUMMARY:
The postpartum period is a critical time for women's physical and psychological health, during which significant hormonal, emotional, and social changes occur. During this period, many women experience increased stress, anxiety, and emotional vulnerability while adapting to new parental responsibilities and caring for a newborn. When these challenges are not adequately managed, they may contribute to the development of postpartum anxiety and postpartum depression, which can negatively affect maternal well-being, mother-infant bonding, breastfeeding practices, and child development. Despite the importance of postpartum mental health, non-pharmacological and easily accessible supportive interventions remain limited.

This randomized controlled experimental study aims to evaluate the effect of a structured, art-based mandala coloring activity on postpartum anxiety and postpartum depression among postpartum women. The study will be conducted at Afyonkarahisar Health Sciences University Health Practice and Research Center, Obstetrics and Gynecology Clinic, and will include women who have recently given birth at this institution. Eligible participants will be randomly assigned to either an intervention group or a control group.

Women in the intervention group will receive individual training in mandala coloring before hospital discharge and will be provided with mandala coloring materials for home use. They will be encouraged to engage in the mandala coloring activity over an eight-week period and will be followed through regular telephone contacts. In addition to monitoring participation in the activity, individualized supportive counseling will be provided based on participants' needs. Women in the control group will receive routine postpartum care without any additional intervention.

Postpartum anxiety and postpartum depression levels will be assessed at multiple time points during the study to examine changes over time. This study seeks to determine whether mandala coloring, as a low-cost and non-pharmacological art-based activity, may serve as a supportive approach to improve psychological well-being during the postpartum period. The findings may contribute to the development of accessible interventions aimed at supporting maternal mental health in the early postpartum period.

DETAILED DESCRIPTION:
The postpartum period begins approximately one hour after delivery and expulsion of the placenta and lasts for six to eight weeks. This period involves not only physiological recovery but also complex psychosocial processes. Changes in parental responsibilities, family dynamics, self-perception, and body image are key components of the postpartum period. The first year after childbirth is considered a particularly sensitive period for women in terms of both physical and psychological health. This sensitivity arises not only from physical recovery but also from the responsibility of caring for a newborn and the effort required to adapt to psychosocial changes.

Because the majority of maternal deaths occur within the first month postpartum and most neonatal deaths occur during the first month of life, the postpartum period is considered a critical time for maternal and newborn health. Stress, anxiety, fatigue, and reduced self-care experienced during this period, when not adequately managed, may increase the risk of postpartum anxiety and postpartum depression. Postpartum depression not only negatively affects maternal physical and mental health but is also associated with early cessation of breastfeeding, impaired mother-infant bonding, delays in child language and behavioral development, disruptions in childhood vaccination schedules, and adverse health outcomes for the entire family. If left untreated, postpartum depression may lead to long-term negative consequences for mothers, children, and families.

The World Health Organization's postpartum care guidelines emphasize the importance of preventive care, counseling services, mental health assessment, family planning, and physical evaluation of both the mother and the infant during the first six weeks postpartum. Counseling topics include breastfeeding, umbilical cord care, emotional well-being, screening for postpartum depression, assessment of domestic violence risk, nutrition, hygiene, safe sexual practices, exercise, iron and folic acid supplementation, and psychosocial support. Despite these recommendations, significant gaps remain in the provision of mental health services during the postpartum transition period, and systematic evaluation of maternal emotional well-being by health professionals is often insufficient. This highlights the need for supportive, non-pharmacological interventions during the postpartum period.

Stress, metabolic changes, and hormonal fluctuations during pregnancy and the postpartum period may increase anxiety levels and contribute to the development of postpartum depression, which is the most common psychiatric disorder following childbirth. Postpartum depression affects not only maternal health but also child development and parenting behaviors. When untreated, it can have profound and lasting negative effects on mothers, children, and families. Early identification of postpartum mental health problems and the implementation of supportive interventions are therefore of critical importance.

Mandala is an art form known to promote psychological relaxation and is typically composed of circular or geometric patterns. Mandalas may be used as a meditation tool and help direct attention to the present moment. Carl Gustav Jung described mandala techniques as therapeutic tools that reflect the individual's inner world and support psychological balance. Mandala practices are generally categorized as unstructured mandalas, which involve free drawing within a circle, and structured mandalas, which involve coloring predefined patterns. Structured mandala coloring is considered an art-based therapeutic approach that enhances attention, mindfulness, and emotional regulation. Although previous studies have demonstrated positive effects of mandala coloring on stress, anxiety, and emotional well-being, research examining its effects on postpartum anxiety and postpartum depression among postpartum women is limited. Therefore, this study aims to investigate the effects of a structured mandala coloring activity on postpartum anxiety and postpartum depression.

This study is designed as a randomized controlled experimental trial and will be conducted at Afyonkarahisar Health Sciences University Health Practice and Research Center, Obstetrics and Gynecology Clinic. The study population will consist of women who give birth at the clinic. Eligible participants will include women who are able to speak and understand Turkish, are 18 years of age or older, are literate, voluntarily agree to participate in the study, and provide written informed consent. Additional inclusion criteria include having no diagnosed psychiatric disorder, not currently receiving psychological or psychiatric support (therapy, counseling, or medication), experiencing no maternal complications during delivery, and having a newborn without congenital malformations, anomalies, or complications. Exclusion criteria include a history of psychological or psychiatric treatment or receiving such treatment during the data collection period, the presence of serious neurological or psychiatric disorders affecting cognitive function, severe health conditions that impair communication or participation in the study, failure to provide informed consent, inability to speak or understand Turkish, and the presence of maternal or neonatal complications during delivery.

Sample size was calculated using G*Power software version 3.1.9.7. Because no previous studies were identified that simultaneously evaluated the effects of mandala art on postpartum anxiety and postpartum depression, effect size estimation was not possible. Therefore, a moderate effect size (f = 0.25), as recommended by Cohen for F-test-based power analysis, was used. The power analysis was conducted with a significance level of α = 0.05 and statistical power of 95% (1-β = 0.95). Based on this analysis, a minimum of 22 participants per group was required. Considering the presence of multiple measurement time points and the time-consuming nature of the data collection process, the sample size was increased to compensate for potential data loss. Accordingly, a total of 60 women, with 30 participants in the intervention group and 30 participants in the control group, were planned to be included in the study.

Participants will be randomized into intervention and control groups using a lottery method. Considering that approximately 30 births occur weekly at the study site, participant selection will be conducted five days per week to prevent scheduling conflicts and ensure feasibility of follow-up. On each recruitment day, women who give birth and meet the inclusion criteria will be assigned to either the intervention or control group. After group allocation, participants will receive detailed information about the study, and the telephone numbers of those who consent to participate will be recorded. Within the hospital setting, only participant selection and mandala training will be conducted, and no additional interventions will be applied.

Participants in the intervention group will receive individual mandala coloring training before hospital discharge. The training will last approximately 20 minutes and will consist of three stages. In the first stage, participants will receive information about mandala coloring. In the second stage, a trained researcher with certification in mandala art will demonstrate the coloring process using a sample mandala. In the third stage, participants will complete a brief practice session on a sample mandala. Following the training, participants will be provided with a mandala coloring set for home use. Participants in the intervention group will be followed for eight weeks, with weekly telephone contacts. During the first contact, a personal information form and the postpartum anxiety and postpartum depression scales will be administered to collect baseline data. In subsequent contacts, the frequency and duration of mandala coloring activities will be assessed, and participants will be asked to share photographs of their completed mandala work via a messaging application.

During telephone follow-ups, individualized counseling will be provided based on participants' needs and questions. Although the counseling will not follow a standardized format, it may include topics such as maternal perineal hygiene, nutrition, breastfeeding, breast care, and basic infant care practices. Postpartum anxiety and postpartum depression scales will be administered at the 1st, 4th, and 8th weeks of the study.

Participants in the control group will not receive any intervention and will continue to receive routine postpartum care. Data from the control group will be collected via telephone at the same time points as the intervention group.

Ethical approval for this study has been obtained. All study procedures will be conducted in accordance with ethical principles governing research involving human participants. Participant confidentiality will be maintained, data will be kept confidential, and participation will be entirely voluntary. Participants will have the right to withdraw from the study at any time without consequences.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish
* Voluntarily agree to participate in the study and have signed the informed consent form
* 18 years of age or older
* Literate
* Have not received any psychiatric diagnosis and are not currently receiving psychological or psychiatric support (therapy, counseling, or medication treatment)
* Have not experienced any complications during delivery
* Have a newborn with no malformation or anomaly
* Have a newborn with no complications

Exclusion Criteria:

* Have previously received psychological or psychiatric treatment or are receiving such treatment during the data collection period,
* Have a serious neurological or psychiatric disorder that affects cognitive functioning,
* Have serious health problems that prevent communication or participation in the study,
* Have not provided informed consent,
* Are unable to speak or understand Turkish,
* Have experienced complications during delivery,
* Have a newborn with a malformation or anomaly,
* Have a newborn with any complications.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is limited to women in the postpartum period who have given birth.
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression | Baseline, week 4, and week 8
  Change in postpartum depression level measured by the Edinburgh Postnatal Depression Scale (EPDS). This scale was developed to determine whether there is a risk of depression in mothers during the postpartum period . The scale consists of 10 items in a four-point Likert format scored between 0 and 3. The minimum score that can be obtained from the scale is 0 and the maximum score is 30. The cut-off score of the scale is 13. Scores above this value indicate a high risk of depression.

SECONDARY OUTCOMES:
Postpartum Anxiety | Baseline, week 4, and week 8
  Change in postpartum anxiety level measured by the Postpartum Anxiety Scale.The original version of the scale was developed and validated with mothers who have infants aged 0-6 months. The scale has the following subdimensions: maternal skills and attachment, newborn well-being and safety, infant care practices, and psychosocial adjustment to motherhood. The maximum possible score that can be obtained from the Likert-type scale is 176, and the cut-off score is 113.5. Higher scores on the scale indicate higher levels of anxiety symptoms.

IPD SHARING:
Plan to Share IPD: No
Individual participant data could be shared in anonymized form; however, no formal data sharing plan has been established for this study.